CLINICAL TRIAL: NCT05471375
Title: Center for Smart Use of Technologies to Assess Real World Outcomes Movement Database
Brief Title: C-STAR Movement Database
Status: Recruiting | Type: Observational
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Arun Jayaraman, PT, PhD, Principal Investigator, Shirley Ryan AbilityLab
Other Study IDs: STU00216350
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Stroke; Parkinson Disease; Lower Limb Amputation Above Knee (Injury); Lower Limb Amputation Below Knee (Injury)
MeSH Terms: conditions — Stroke; Parkinson Disease; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Stroke: For this cohort, individuals who have experienced a stroke will be asked to complete a variety of movement related rehabilitation assessments with wearable sensors and audio/video recording.
  Interventions: Other: Database Entry
- Parkinsons Disease: For this cohort, individuals who have been diagnosed with Parkinsons Disease will be asked to complete a variety of movement related rehabilitation assessments with wearable sensors and audio/video recording.
  Interventions: Other: Database Entry
- Lower Limb Amputation: For this cohort, individuals who have experienced a lower limb amputation will be asked to complete a variety of movement related rehabilitation assessments with wearable sensors and audio/video recording.
  Interventions: Other: Database Entry
- Healthy Control: For this cohort, individuals who have no significant neurologic or orthopedic injuries will be asked to complete a variety of movement related rehabilitation assessments with wearable sensors and audio/video recording.
  Interventions: Other: Database Entry

INTERVENTIONS:
Other: Database Entry — Database entries will contain wearable sensor, audio, and video data collected during rehabilitation-related movement assessments

SUMMARY:
The purpose of this study is to develop a database that contains movement and rehabilitation-related data collected through the use of wearable sensors and video. This database will serve as a resource for clinicians and researchers interested in the investigation of movement or rehabilitation-related research ideas.

DETAILED DESCRIPTION:
Scholarly research in the field of physical rehabilitation helps to aid in maximizing outcomes for individuals that require these services due to orthopedic and neurologic injuries. To produce quality research results, large cohorts of individuals are often required for data analysis. Some research facilities or labs do not have adequate access to large cohorts or may not have the means to recruit them. By building the C-STAR database, the intent is to create a database that can serve as a hub for data sets that researchers and clinicians with appropriate access may use to support their research questions related to movement and physical rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 0 to 99 years old
2. Able and willing to give written consent and comply with study procedures

Exclusion Criteria:

1. Unable to give written consent or comply with study procedures
2. Any condition that would prevent safe completion of study activities, as determined by the Principal Investigator

Max Age: 99 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: By building the C-STAR database, the intent is to create a database that can serve as a hub for data sets that researchers and clinicians with appropriate access may use to support their research questions related to movement and physical rehabilitation.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-08-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Database development | Data will be collected and added to the C-STAR database for 3 years
  To develop an online database that contains movement and rehabilitation-related data collected with wearable sensors and video that may be accessed, with appropriate permissions, by clinicians and researchers that are interested in the investigation of movement or rehabilitation related research ideas.

CONTACTS AND LOCATIONS:
Overall Officials: Arun Jayaraman, PT, PhD, Principal Investigator — Shirley Ryan AbilityLab; Levi Hargrove, PhD, Principal Investigator — Shirley Ryan AbilityLab; Richard Lieber, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States